CLINICAL TRIAL: NCT01582685
Title: Exercise in Breast Cancer Survivors: Analysis of Angiogenic Profile
Brief Title: Exercise in Breast Cancer Survivors
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no patients enrolled
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, Natale Sheehan, Assistant Professor of Medicine, University of Mississippi Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2011-0121
Record Dates: First submitted 2012-04-02; First posted 2012-04-23 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Breast Cancer; Obesity
Keywords: Breast Cancer; Obesity; Exercise; Angiogenesis
MeSH Terms: conditions — Breast Neoplasms; Obesity; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise Group (Experimental): The intervention is a structured walking program which will be performed partly in the Pavilion Physical Therapy clinic and partly at home. The participant will be instructed in how hard to exercise, how long to exercise, and how many times in a week to exercise. You will also be instructed in how to exercise safely.
  Interventions: Behavioral: Exercise
- No Exercise (No Intervention): These participants will receive standard of care follow up.

INTERVENTIONS:
Behavioral: Exercise — The participant will exercise for 16 weeks under supervision. The exercise regimen is increased slowly over 16 weeks.
  Arms: Exercise Group

SUMMARY:
The investigators hypothesize that exercise in postmenopausal breast cancer survivors will result in an increase in the plasma concentrations of angiostatic factors and a decrease in the plasma concentrations of angiogenic factors. Exercise is expected to result in a circulating angiostatic phenotype that inhibits adipose tissue mass, growth of breast cancer tumor, growth of microscopic residual disease after breast cancer resection, decreases rates of local-regional recurrence, decreases rates of distant recurrence, and increases survival.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age and < 65 years of age
* Female
* BMI > 25
* Weight < 350 pounds
* English as a primary language
* Postmenopausal
* Invasive ER-positive cancer on biopsy and subsequent definitive surgical therapy
* Received and Completed standard of care adjuvant therapy (Concurrent endocrine therapy acceptable)
* 6-12 months after completion of therapy (excluding adjuvant endocrine therapy) at time of randomization

Exclusion Criteria:

* Recurrent breast cancer
* DCIS only (no invasive component)
* Taking a Beta Blocker or Verapamil
* Pregnant
* Wheelchair bound
* Unable to ambulate independently
* Concurrent uncontrolled medical or psychiatric disorder
* Open wound
* Stage IV breast cancer
* Progression of disease
* Bilateral mastectomies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Number of participants that complete the study as a measure of feasibility of an exercise intervention in obese breast cancer survivors. | 12 months
  Number of participants that enroll in the study and actually complete the study

SECONDARY OUTCOMES:
IGF-1, endostatin, and VEGF levels in obese breast cancer survivors undergoing an exercise intervention as a measure of angiostatic phenotype: | 12 months
  IFG-1 levels,unbound VEGF levels, Endostatin levels
Amount of adipose tissue mass as measured on CT scans in obese breast cancer survivors before and after exercise intervention as a measure of weight loss | 12 months
  Adipose tissue mass volume as measured on CT scan

CONTACTS AND LOCATIONS:
Overall Officials: Natale Sheehan, MD, Principal Investigator — University of Mississippi Health Care
Locations (1):
- University of Mississippi Health Care, Jackson, Mississippi, United States